CLINICAL TRIAL: NCT04924829
Title: Safety and Effectiveness Observational Study of Anti IL-6 Tocilizumab in Hospital Admitted Patients With Severe COVID-19 Pneumonia.
Brief Title: Safety and Effectiveness Study of Tocilizumab in Patients With Severe COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, ANACLARA MURUJOSA, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 6052
Record Dates: First submitted 2021-06-10; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Severe COVID 19 Pneumonia; Tocilizumab
Keywords: covid 19; tocilizumab; severe pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tocilizumab: Group that received tocilizumab (8mg/kg, maximum dose 800 mg, only once) while being admitted with severe COVID-19 pneumonia.
  Interventions: Drug: Tocilizumab
- Non-tocilizumab: Group that did not receive tocilizumab but share the same indication according to the elegibility criteria for it as the tocilizumab group while admitted with severe COVID-19 pneumonia.

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab received as a single intravenous infusion over the period of 60 minutes. Dose of 8 mg/kg, maximum dose of 800 mg.
  Groups: Tocilizumab

SUMMARY:
Retrospective observational cohort study to evaluate the safety and effectiveness of tocilizumab in the treatment of severe COVID-19 pneumonia

DETAILED DESCRIPTION:
Since the appearence of the disease today known as COVID-19 there has been multiple interventions to try to gain knowledge on the subject and obtain a benefitial effect treating this condition.

Tocilizumab, a monoclonal antibody targeting IL-6 receptor has arised as an alternative for the treament of COVID-19 pneumonia.

It is a drug used for the treatment of rhemautoid arthritis and other autoimmune diseases as well as approved in recent years for the treatment of the cytokine release syndrome (CRS) in CAR-T therapy.

It is based in this last premise that the benefitial effect on COVID-19 pneumonia has been sought of. According to investigation into the physiopathology of the virus, it is supposed to trigger the inflamattory cascade that generates damage to lungs and creates the most severe cases of the disease. These findings could imply that tocilizumab may serve to interrupt this cytokine storm and prevent the progression of the disease.

The aim of the study is to evaluate the effectiveness and safety of tocilizumab in the treatment of severe cases of COVID-19. For that purpose, an observational retrospective cohort study has been designed comparing two populations that share the same indication for the treatment with tocilizumab. One having received the drug and the other in a close previous period of time that has not received it because of lack of availability or generalisation of its use. Mortality will be assesed as well as other variables such as need for mechanical ventilation and adverse effects of tocilizumab.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admitted patients with severe COVID-19 pneumonia (Individuals who have SpO2 <94% on room air at sea level, a ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) <300 mm Hg, respiratory frequency >30 breaths/min, or lung infiltrates >50%).
* Confirmed diagnosis of Covid-19 through qualitative polymerase-reverse transcriptase (qRT-PCR -GeneDX Co, Ltd o similar) or antigen rapid test.
* Patients who received tocilizumab or shared the same indication but did not received it (same period of time or previous close period) that:

  * Progress in the requirement of supplemental oxygen (over 3L/m) and/or use of non-rebreathing mask with 8L/m or more to mantain a Sp02>= 94%.

AND

* Active inflammatory state defined as persistent fever > 38°C (defined as 2 or more measurements in a 24-hour period from hospital admission) despite the use of dexamethasone in the previous 48 hours OR C reactive Protein > 50 mg /dL OR D Dimer > 1000 ng/mL.

Exclusion Criteria:

* Asymptomatic, mild or moderate COVID-19 disease.
* Patients with some type of immunosupression (HIV, use of immunomodulatory drugs, organ-trasplant receipt patients)
* Pregnant or breast-feeding
* Patients with augmented risk of bowel perforation (history of diverticulitis or bowel surgery in the three months prior to the study entrance date)
* Known severe allergic reactions to TCZ
* Suspected active bacterial, fungal, viral, or other infection (besides COVID-19)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 x upper limit of normal (ULN) at screening
* Absolute neutrophil count (ANC) < 1000/mL at screening
* Platelet count < 50,000/mL at screening
* Positive Hepatitis B Surface (HbS) antigen
* Procalcitonine > 0,5 ng/mL
* Day of symptom onset before day 7 or after day 12
* Patients with dementia
* Patients non eligible to progress to mechanical ventilation because of frailty/comorbidites according to medical decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital with severe COVID-19 pneumonia that have progressed in the requirement of oxygen or need of non-rebreathing mask that have an active inflammatory state defined as persistent fever, CRP over 50 mg/dL or D dimer over 1000 ng/dL.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days from hospital admission
  28-day mortality
Percentage of patients in invasive mechanical ventilation at day 28 | 28 days from hospital admission
  Percentage of patients that received invasive mechanical ventilation at day 28 following hospital admission.
Clinical status during follow-up at 28th day | 28th day from hospital admission
  Ordinal outcome with seven mutually exclusive categories to describe the patient's clinical status during follow-up. The six categories are: (1) Discharged or ready for discharge; (2) Admitted to non-ICU ward without oxygen; (3) admitted to non-ICU ward but requiring supplemental oxygen; (4) admitted to ICU or non ICU ward requiring high flow nasal canula or other non invasive mechanical ventilation; (5) admitted to ICU ward requiring invasive mechanical ventilation (6) admitted to ICU ward requiring extracorporeal membrane oxygenation or invasive mechanical ventilation plus other vital organ support; (7) death

SECONDARY OUTCOMES:
Mortality rate | Days 14 and 21
Percentage of patients in invasive mechanical ventilation at day 14 and 21 | Days 14 and 21
Percentage of patients with hospital discharge at day 7, 14, 21 and 28 | Days 7, 14, 21 and 28
Time to hospital discharge | Up to 60 days
  Time from hospital admission to hospital discharge
Percentage of patients admitted to ICU-ward at day 28 | 28th day from hospital admission
  Percentage of patients admitted to ICU-ward at day 28 from hospital admission
Time to Improvement of at Least 2 Categories Relative to Baseline on a 7-Category Ordinal Scale of Clinical Status | Up to 60 days
Percentage of patients with need of tracheostomy at day 28 of hospital admission | 28th day from hospital admission
Time to mechanical ventilation from hospital admission | Up to 28 days
Days of ICU admission | Up to 60 days
Time to ICU discharge from hospital admission | Up to 60 days
  Time to ICU discharge from hospital admission in the patients subgroup that required ICU admission.
Percentage of patients with adverse effects / serious adverse effects | Up to 28 days
Percentage of superimposed infections | 28th day from hospital admission

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos AIres, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] RECOVERY Collaborative Group; Horby P, Lim WS, Emberson JR, Mafham M, Bell JL, Linsell L, Staplin N, Brightling C, Ustianowski A, Elmahi E, Prudon B, Green C, Felton T, Chadwick D, Rege K, Fegan C, Chappell LC, Faust SN, Jaki T, Jeffery K, Montgomery A, Rowan K, Juszczak E, Baillie JK, Haynes R, Landray MJ. Dexamethasone in Hospitalized Patients with Covid-19. N Engl J Med. 2021 Feb 25;384(8):693-704. doi: 10.1056/NEJMoa2021436. Epub 2020 Jul 17. PMID 32678530
- [Background] Rubbert-Roth A, Furst DE, Nebesky JM, Jin A, Berber E. A Review of Recent Advances Using Tocilizumab in the Treatment of Rheumatic Diseases. Rheumatol Ther. 2018 Jun;5(1):21-42. doi: 10.1007/s40744-018-0102-x. Epub 2018 Mar 3. PMID 29502236
- [Background] Zhu J, Pang J, Ji P, Zhong Z, Li H, Li B, Zhang J. Elevated interleukin-6 is associated with severity of COVID-19: A meta-analysis. J Med Virol. 2021 Jan;93(1):35-37. doi: 10.1002/jmv.26085. Epub 2020 Oct 30. No abstract available. PMID 32470146
- [Background] Stone JH, Frigault MJ, Serling-Boyd NJ, Fernandes AD, Harvey L, Foulkes AS, Horick NK, Healy BC, Shah R, Bensaci AM, Woolley AE, Nikiforow S, Lin N, Sagar M, Schrager H, Huckins DS, Axelrod M, Pincus MD, Fleisher J, Sacks CA, Dougan M, North CM, Halvorsen YD, Thurber TK, Dagher Z, Scherer A, Wallwork RS, Kim AY, Schoenfeld S, Sen P, Neilan TG, Perugino CA, Unizony SH, Collier DS, Matza MA, Yinh JM, Bowman KA, Meyerowitz E, Zafar A, Drobni ZD, Bolster MB, Kohler M, D'Silva KM, Dau J, Lockwood MM, Cubbison C, Weber BN, Mansour MK; BACC Bay Tocilizumab Trial Investigators. Efficacy of Tocilizumab in Patients Hospitalized with Covid-19. N Engl J Med. 2020 Dec 10;383(24):2333-2344. doi: 10.1056/NEJMoa2028836. Epub 2020 Oct 21. PMID 33085857
- [Background] RECOVERY Collaborative Group. Tocilizumab in patients admitted to hospital with COVID-19 (RECOVERY): a randomised, controlled, open-label, platform trial. Lancet. 2021 May 1;397(10285):1637-1645. doi: 10.1016/S0140-6736(21)00676-0. PMID 33933206
- [Background] REMAP-CAP Investigators; Gordon AC, Mouncey PR, Al-Beidh F, Rowan KM, Nichol AD, Arabi YM, Annane D, Beane A, van Bentum-Puijk W, Berry LR, Bhimani Z, Bonten MJM, Bradbury CA, Brunkhorst FM, Buzgau A, Cheng AC, Detry MA, Duffy EJ, Estcourt LJ, Fitzgerald M, Goossens H, Haniffa R, Higgins AM, Hills TE, Horvat CM, Lamontagne F, Lawler PR, Leavis HL, Linstrum KM, Litton E, Lorenzi E, Marshall JC, Mayr FB, McAuley DF, McGlothlin A, McGuinness SP, McVerry BJ, Montgomery SK, Morpeth SC, Murthy S, Orr K, Parke RL, Parker JC, Patanwala AE, Pettila V, Rademaker E, Santos MS, Saunders CT, Seymour CW, Shankar-Hari M, Sligl WI, Turgeon AF, Turner AM, van de Veerdonk FL, Zarychanski R, Green C, Lewis RJ, Angus DC, McArthur CJ, Berry S, Webb SA, Derde LPG. Interleukin-6 Receptor Antagonists in Critically Ill Patients with Covid-19. N Engl J Med. 2021 Apr 22;384(16):1491-1502. doi: 10.1056/NEJMoa2100433. Epub 2021 Feb 25. PMID 33631065
- [Background] Angriman F, Ferreyro BL, Burry L, Fan E, Ferguson ND, Husain S, Keshavjee SH, Lupia E, Munshi L, Renzi S, Ubaldo OGV, Rochwerg B, Del Sorbo L. Interleukin-6 receptor blockade in patients with COVID-19: placing clinical trials into context. Lancet Respir Med. 2021 Jun;9(6):655-664. doi: 10.1016/S2213-2600(21)00139-9. Epub 2021 Apr 27. PMID 33930329
- [Background] McCreary EK, Angus DC. Efficacy of Remdesivir in COVID-19. JAMA. 2020 Sep 15;324(11):1041-1042. doi: 10.1001/jama.2020.16337. No abstract available. PMID 32821934
- [Background] Zhang X, Peck R. Clinical pharmacology of tocilizumab for the treatment of patients with rheumatoid arthritis. Expert Rev Clin Pharmacol. 2011 Sep;4(5):539-58. doi: 10.1586/ecp.11.33. PMID 22114882
- [Background] Pons S, Fodil S, Azoulay E, Zafrani L. The vascular endothelium: the cornerstone of organ dysfunction in severe SARS-CoV-2 infection. Crit Care. 2020 Jun 16;24(1):353. doi: 10.1186/s13054-020-03062-7. PMID 32546188
- [Background] Hermine O, Mariette X, Tharaux PL, Resche-Rigon M, Porcher R, Ravaud P; CORIMUNO-19 Collaborative Group. Effect of Tocilizumab vs Usual Care in Adults Hospitalized With COVID-19 and Moderate or Severe Pneumonia: A Randomized Clinical Trial. JAMA Intern Med. 2021 Jan 1;181(1):32-40. doi: 10.1001/jamainternmed.2020.6820. PMID 33080017
- [Background] Salvarani C, Dolci G, Massari M, Merlo DF, Cavuto S, Savoldi L, Bruzzi P, Boni F, Braglia L, Turra C, Ballerini PF, Sciascia R, Zammarchi L, Para O, Scotton PG, Inojosa WO, Ravagnani V, Salerno ND, Sainaghi PP, Brignone A, Codeluppi M, Teopompi E, Milesi M, Bertomoro P, Claudio N, Salio M, Falcone M, Cenderello G, Donghi L, Del Bono V, Colombelli PL, Angheben A, Passaro A, Secondo G, Pascale R, Piazza I, Facciolongo N, Costantini M; RCT-TCZ-COVID-19 Study Group. Effect of Tocilizumab vs Standard Care on Clinical Worsening in Patients Hospitalized With COVID-19 Pneumonia: A Randomized Clinical Trial. JAMA Intern Med. 2021 Jan 1;181(1):24-31. doi: 10.1001/jamainternmed.2020.6615. PMID 33080005
- [Background] Veiga VC, Prats JAGG, Farias DLC, Rosa RG, Dourado LK, Zampieri FG, Machado FR, Lopes RD, Berwanger O, Azevedo LCP, Avezum A, Lisboa TC, Rojas SSO, Coelho JC, Leite RT, Carvalho JC, Andrade LEC, Sandes AF, Pintao MCT, Castro CG Jr, Santos SV, de Almeida TML, Costa AN, Gebara OCE, de Freitas FGR, Pacheco ES, Machado DJB, Martin J, Conceicao FG, Siqueira SRR, Damiani LP, Ishihara LM, Schneider D, de Souza D, Cavalcanti AB, Scheinberg P; Coalition covid-19 Brazil VI Investigators. Effect of tocilizumab on clinical outcomes at 15 days in patients with severe or critical coronavirus disease 2019: randomised controlled trial. BMJ. 2021 Jan 20;372:n84. doi: 10.1136/bmj.n84. PMID 33472855
- [Background] Salama C, Han J, Yau L, Reiss WG, Kramer B, Neidhart JD, Criner GJ, Kaplan-Lewis E, Baden R, Pandit L, Cameron ML, Garcia-Diaz J, Chavez V, Mekebeb-Reuter M, Lima de Menezes F, Shah R, Gonzalez-Lara MF, Assman B, Freedman J, Mohan SV. Tocilizumab in Patients Hospitalized with Covid-19 Pneumonia. N Engl J Med. 2021 Jan 7;384(1):20-30. doi: 10.1056/NEJMoa2030340. Epub 2020 Dec 17. PMID 33332779
- [Background] Soin AS, Kumar K, Choudhary NS, Sharma P, Mehta Y, Kataria S, Govil D, Deswal V, Chaudhry D, Singh PK, Gupta A, Agarwal V, Kumar S, Sangle SA, Chawla R, Narreddy S, Pandit R, Mishra V, Goel M, Ramanan AV. Tocilizumab plus standard care versus standard care in patients in India with moderate to severe COVID-19-associated cytokine release syndrome (COVINTOC): an open-label, multicentre, randomised, controlled, phase 3 trial. Lancet Respir Med. 2021 May;9(5):511-521. doi: 10.1016/S2213-2600(21)00081-3. Epub 2021 Mar 4. PMID 33676589
- See also: WHO Coronavirus (COVID-19) Dashboard — https://covid19.who.int/
- See also: A minimal common outcome measure set for COVID-19 clinical research — https://doi.org/10.1016/S1473-3099(20)30483-7
- See also: Ordered Logistic Regression | Stata Annotated Output — https://stats.idre.ucla.edu/stata/output/ordered-logistic-regression/
- See also: Brant R. Assessing proportionality in the proportional odds model for ordinal logistic regression. Biometrics [Internet]. 1990 Dec;46(4):1171-8. — https://www.ncbi.nlm.nih.gov/pubmed/2085632
- See also: Ho DE, Imai K, King G, Stuart EA. Matching as Nonparametric Preprocessing for Reducing Model Dependence in Parametric Causal Inference [Internet]. Vol. 15, Political Analysis. 2007. p. 199-236. — http://dx.doi.org/10.1093/pan/mpl013
- See also: Matschinger H, Heider D, König H-H. A Comparison of Matching and Weighting Methods for Causal Inference Based on Routine Health Insurance Data, or: What to do If an RCT is Impossible. Gesundheitswesen [Internet]. 2020 Mar;82(S 02):S139-50. — http://dx.doi.org/10.1055/a-1009-6634
- See also: ACTUALIZACIONES BASADAS EN EVIDENCIA COVID-19 Tocilizumab para el tratamiento de pacientes con COVID-19 — https://www.argentina.gob.ar/sites/default/files/informe-covid-19-n6-tocilizumab.pdf
- See also: IDS COVID 19 guideline treatment and management — https://www.idsociety.org/practice-guideline/covid-19-guideline-treatment-and-management/